CLINICAL TRIAL: NCT04247763
Title: Fast Food, Fatigue, and Inflammation: The FOOD Study
Brief Title: Fast Food, Fatigue, and Inflammation
Acronym: FOOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Janice Kiecolt-Glaser, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: OSU-10078; NCI-2014-01312 (Registry Identifier: CTRP)
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized crossover trial: participants were randomized to sequence of meal type; they ate one high saturated fat meal and one high oleic sunflower oil meal with 1-4 weeks washout in between meals
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind: The data manager assigned arbitrary names to each meal so that only the data manager and the kitchen staff were unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Saturated Fat Meal, Oleic Sunflower Oil Meal) (Experimental)
  Interventions: Other: Saturated Fat Meal; Other: Oleic Sunflower Oil Meal
- Arm 2 (Oleic Sunflower Oil Meal, Saturated Fat Meal) (Active Comparator)
  Interventions: Other: Saturated Fat Meal; Other: Oleic Sunflower Oil Meal

INTERVENTIONS:
Other: Saturated Fat Meal
Other: Oleic Sunflower Oil Meal

SUMMARY:
This double-blind, randomized crossover trial assessed inflammation and fatigue following a fast-food-type meal (saturated fat) compared to a healthier meal (monounsaturated fat) in breast cancer survivors and benign controls (women who had an initial abnormal test for breast cancer).

ELIGIBILITY:
Inclusion Criteria:

* We recruited a subset of a larger parent longitudinal observational study to participate in this study. Initially, participants were recruited following an abnormal mammogram, which resulted in either a malignant (cancer group) or benign (non-cancer control group) diagnosis.

Exclusion Criteria:

* A history of any prior cancer except basal or squamous cell, chronic obstructive pulmonary disease, evidence of liver or kidney failure, symptomatic ischemic heart disease, significant visual or auditory problems, cognitive impairment, major medical conditions involving the immune system such as diabetes, autoimmune and/or inflammatory diseases including rheumatoid arthritis and ulcerative colitis, alcohol or drug abuse, marked and recurrent gastrointestinal problems, or regular use of medications with major immunological consequences, e.g., steroids.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-12-13 (Actual); Primary Completion 2013-06-11 (Actual); Study Completion 2013-06-11 (Actual)

PRIMARY OUTCOMES:
Post-Meal Change in C-reactive Protein | Blood samples were obtained before the meal (baseline) as well as 2, 4, and 7 hours post-meal
  Serum CRP was obtained from blood drawn before the meal as well as 2, 4, and 7 hours post-meal. It was measured with the Vascular Injury Panel 2 Multispot Kit on an MSD Imager 2400 (both Meso Scale Discovery, Rockville, MD, USA), following kit instructions.
Post-Meal Change in Serum Amyloid A | Blood samples were obtained before the meal (baseline) as well as 2, 4, and 7 hours post-meal
  Serum Amyloid A was obtained from blood drawn before the meal as well as 2, 4, and 7 hours post-meal. It as measured with the Vascular Injury Panel 2 Multispot Kit on an MSD Imager 2400 (both Meso Scale Discovery, Rockville, MD, USA), following kit instructions.
Change in Intercellular adhesion molecule-1 | Blood samples were obtained before the meal (baseline) as well as 2, 4, and 7 hours post-meal
  sICAM-1 was obtained from blood drawn before the meal as well as 2, 4, and 7 hours post-meal. It was measured with the Vascular Injury Panel 2 Multispot Kit on an MSD Imager 2400 (both Meso Scale Discovery, Rockville, MD, USA), following kit instructions.
Change in Vascular cell adhesion molecule-1 | Blood samples were obtained before the meal (baseline) as well as 2, 4, and 7 hours post-meal
  sVCAM-1 was obtained from blood drawn before the meal as well as 2, 4, and 7 hours post-meal. It was measured with the Vascular Injury Panel 2 Multispot Kit on an MSD Imager 2400 (both Meso Scale Discovery, Rockville, MD, USA), following kit instructions.
Fatigue at Follow-Up Visits | The survey was administered upon admission to the Clinical Research Center before the meal at both visits and at 18- and 30-month follow-up visits.
  The 30-item Multidimensional Fatigue Symptom Inventory-Short form assesses behavioral, cognitive, physical, and affective expressions of fatigue. It provides a very good measure of the multidimensional aspects of fatigue, allows for comparisons between fatigued and non-fatigued individuals, and has subscales measuring general, physical, emotional, mental, and vigor aspects of fatigue, as well as a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Kiecolt-Glaser, Principal Investigator — Ohio State Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madison AA, Belury MA, Andridge R, Shrout MR, Renna ME, Malarkey WB, Bailey MT, Kiecolt-Glaser JK. Afternoon distraction: a high-saturated-fat meal and endotoxemia impact postmeal attention in a randomized crossover trial. Am J Clin Nutr. 2020 Jun 1;111(6):1150-1158. doi: 10.1093/ajcn/nqaa085. PMID 32393980
- See also: Related Info — http://cancer.osu.edu